CLINICAL TRIAL: NCT03288701
Title: SCALE HF - Smart SCALEs With Bioelectrical Impedance Analysis for Treatment Guidance in Decompensated Heart Failure
Brief Title: Smart SCALEs With Bioimpedance Analysis for Treatment Guidance in Decompensated Heart Failure
Acronym: SCALE HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 2017-00845
Record Dates: First submitted 2017-07-25; First posted 2017-09-20 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; With Decompensation
Keywords: heart failure; cardial decompensation; smart scale; bioimpedance analysis; whole body water
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Composition Analysis (Experimental): Daily measurement of the Body Composition using electrical Bioimpedance Analysis in a scale (seca mBCA 515). Including total body water and weight.
  Interventions: Device: Seca medical Body Composition Analyser 515

INTERVENTIONS:
Device: Seca medical Body Composition Analyser 515 — Comparison of reduction of whole body water and body weight in patients with decompensated heart failure under forced diuretic treatment

SUMMARY:
In this trial the measurement of whole body water will be compared to the standard method of measuring the body weight as treatment guidance in patients with decompensated heart failure. The Seca mBCA 515 [medical Body Composition Analyser] will be used to quantify the whole body water by using bioelectrical impedance analysis.

DETAILED DESCRIPTION:
Investigators will include 153 participants hospitalized in the University Hospital in Basel. Daily measurements of whole body water and body weight will be performed in each person until diuretic treatment is stopped or the patient is discharged from hospital, respectively.

Primary endpoint is the correlation between reduction of whole body water (in kg) and reduction of body weight (in kg) in patients with decompensated heart failure receiving forced diuretic treatment (max. deviation +/- 1kg).

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* hospitalization because of decompensated heart failure treated with forced diuresis
* able to stand on the scale without help from others and able to hold handrails with both hands

Exclusion Criteria:

* refusal to share personal data
* implantable electronic device (e.g. Pacemaker, etc.)
* condition that does not allow skin contact of soles of feet and scale or hands with handrail (leg prosthesis, wounds, bandage, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Measurement of total body water (TBW) in kg | From baseline until the date of hospital discharge or stop date of forced diuretic treatment, whichever came first, assessed up to 2 weeks.
  total body water (TBW) in kg will be measured daily
Measurement of body weight (BW) in kg | From baseline until the date of hospital discharge or stop date of forced diuretic treatment, whichever came first, assessed up to 2 weeks.
  body weight (BW) in kg will be measured daily

SECONDARY OUTCOMES:
Measurement of fatty tissue (FT) in kg | From baseline until the date of hospital discharge or stop date of forced diuretic treatment, whichever came first, assessed up to 2 weeks.
  To provide a more exact comparison of total body water and body weight, fatty mass will be subtracted from the body weight. Subsequently the absolute difference between the reduction of the total body water (in kg) and the reduction of the body weight (in kg), in which fatty tissue (in kg) was subtracted, will be calculated (e.g. (BW day 1- FT day 1) - (BW day 2 - FT day 2) = reduction of BW without fatty tissue).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No